CLINICAL TRIAL: NCT01956292
Title: Observational Study of Continous Monitoring of Arterial Blood Pressure in Spontaneous Intraparenchimal Cerebral Haemorrhage
Brief Title: Continuous Monitoring of Blood Pressure in Spontaneous Intraparenchimal Cerebral Haemorrhage
Acronym: BP-MONICH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Sant'Anna (Other)
Responsible Party: Principal Investigator, Simone Vidale, M.D., Azienda Ospedaliera Sant'Anna
Other Study IDs: OSA-0002
Record Dates: First submitted 2013-09-29; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Intraparenchimal Cerebral Haemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intraparenchimal cerebral haemorrhage

SUMMARY:
Evaluation of blood pressure variability in the acute phase of intraparenchimal cerebral haemorrhage and its consequences to clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* hospitalization only for spontaneous intraparenchimal cerebral haemorrhage
* age over 18 years

Exclusion Criteria:

* cerebral haemorrhage secondary to other causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital for intraparenchimal cerebral haemorrhage
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
evaluation of blood pressure varibility on clinical course in patients with cerebral haemorrhage | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- AO Sant'Anna Hospital, Como, Como, Italy